CLINICAL TRIAL: NCT06826521
Title: Radiological and Functional Outcomes of Internal Fixation Methods for Ipsilateral Femoral Neck and Shaft Fractures in Young Adult Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Ibrahim khalifa yakoup, Principal investigator (Orthopedic resident at orthopedic and trauma surgery department at Assiut university hospitals ), Assiut University
Other Study IDs: RFOIFMIFNSFYAP
Record Dates: First submitted 2025-01-31; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Ipsilateral Neck and Shaft Fractures and Internal Fixation Method and Follow Up At One Year Postoperative for Radiological and Functional Outcomes
Keywords: Radiological and functional outcomes of internal fixation methods for ipsilateral femoral neck and shaft fractures in young adult patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- I will compare results with favourable outcomes between single and dual constructs
  Interventions: Procedure: Single construct versus dual constructs will give satisfactory radiological and functional outcomes

INTERVENTIONS:
Procedure: Single construct versus dual constructs will give satisfactory radiological and functional outcomes — Single construct like cephalomedullary nail or long DHS in fixation of both neck and shaft fractures, dual constructs like DHS or cannulated screws and retrograde nail or DHS or cannulated screws and dymanic compression plate in fixation of both fractures.

SUMMARY:
Does the single construct produce more favourable radiological and functional outcomes with less complication when it is compared to dual constructs for fixation of ipsilateral femoral neck and shaft fractures in young adult patients at one year follow up?

DETAILED DESCRIPTION:
The investigators will do follow up for internal fixation methods for ipsilateral femoral neck and shaft fractures in young adult patients at one year and observe does single construct will give favourable outcomes versus dual constructs?

ELIGIBILITY:
Inclusion Criteria:

* Age of the patients from 18 to 55 years
* Recent fracture within one week
* Ipsilateral Neck and shaft femur fractures according to AO Classification including 31 B (all types of neck ) and 32 A,B and C ( all types of shaft femur )

Exclusion Criteria:

* Open fractures GIII
* patients more than 55 and less than 18 years old
* Patient with comorbidities: uncontrolled D.M, renal patient, neurological deficits.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adult patients from 18- 55 years old not more than and not less Not with comrbodities like uncontrolled diabetes,renal disease and neurological deficits.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Radiological union evaluation | Assessment of radiological union and the time will be taken at one year follow up
  Radiographic union evaluation of ipsilateral neck and shaft femur fractures after internal fixation methods at one year follow up in young adult patients using :
  Radiographic union score of the hip for neck fracture Radiographic union score for the femur fracture. Minimum score for these scales is 10 and maximum is 30 High score means good outcome

SECONDARY OUTCOMES:
Functional outcome | One year follow up
  Functional outcome will be assessed after internal fixation methods for ipsilateral femoral neck and shaft fractures in young adult patients using friedman and wyman scale to assess whether patients have pain , Impaired daily life activities and loss of hip and knee range of motion . this scale is categorised by good, fair and poor outcome Good which have no pain no impaired daily life activities and less than 20 % loss of hip and knee range of motion Fair mild impaired daily life activities, mild to moderate pain and 20_50% loss of hip and knee range of motion Poor moderate impaired daily life activities, severe pain and more than 50% loss of hip and knee range of motion.
Complications | One year follow up
  Complications will be reported if occured like non- union, infection and avascular necrosis of the neck.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://journals.lww.com/jorthotrauma/fulltext/2008/02000/Functional_Outcome_of_Ipsilateral.00005.aspx